CLINICAL TRIAL: NCT02190435
Title: Computer-Assisted Navigation for Intramedullary Nail Fixation of Intertrochanteric Femur Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Collaborators: Stryker Orthopaedics (Industry)
Responsible Party: Principal Investigator, Kevin Grant, MD, Principal Investigator, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-111
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-04

CONDITIONS: Intertrochanteric Femur Fractures
Keywords: Computer-assisted navigation; ADAPT; Intramedullary nail; Intertrochanteric femur fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- ADAPT (Experimental): Patients that receive intramedullary nail fixation with use of the Stryker ADAPT computer-assisted navigation system
  Interventions: Device: Stryker ADAPT computer-assisted navigation
- Control (Active Comparator): Patients that receive conventional technique intramedullary nail fixation without use of the Stryker ADAPT computer-assisted navigation system
  Interventions: Device: Conventional technique

INTERVENTIONS:
Device: Stryker ADAPT computer-assisted navigation — Adaptive Positioning Technology for Gamma 3
  Arms: ADAPT
Device: Conventional technique — Conventional Technique
  Arms: Control

SUMMARY:
There are approximately 250,000 hip fractures in the US every year, and intertrochanteric (IT) fractures (fractures that occur just below the femoral head) account for nearly half of these fractures. The use of intramedullary (IM) nails for fixation of IT femur fractures has become a well-accepted and increasingly more common procedure among orthopaedic traumatologists, and is standard of care at our institution.

While advancements in intramedullary nail fixation have made it a relatively efficient procedure, the placement of the lag screw into the femoral head still remains a challenging step in the procedure. Inaccurate placement can lead to screw cut-out, one of the most commonly reported complications with IM nail fixation. Previous work has shown that the lag screw position is an important factor in reducing screw cut-out. This step of the procedure can be time demanding and often requires several intraoperative radiographs for accurate placement. Recently developed computer-assisted navigation systems provide surgeons with the ability to track screw placement in real-time. This could allow for improved screw placement and potentially reduce radiation exposure to the patient and surgeon. To date, the potential advantages of computer-assisted navigation have not been examined.

The primary objective of this study is to examine whether the use of Stryker's ADAPT computer-assisted navigation for Gamma nail fixation can result in improved lag screw placement. The secondary objective is to examine whether the use of the ADAPT for Gamma nail fixation can reduce intraoperative radiation exposure.Our hypothesis is that there is a difference in the lag screw placement (i.e. tip to apex distance measurement) between procedures using the ADAPT system versus the conventional technique for Gamma nail fixation. Additionally, we hypothesize that there is a difference in radiation exposure (i.e. fluoroscopy time) between procedures using the ADAPT system versus the conventional technique for Gamma nail fixation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hip fracture fixation with a Gamma Nail by one of four orthopaedic trauma surgeons at William Beaumont Hospital Royal Oak
* Diagnosis of an intertrochanteric femur fracture (AO Classification 31-A1,A2)
* Low energy mechanism of injury (i.e. fall, twist)

Exclusion Criteria:

* Minors (less than 18 years)
* Pregnant
* Have a high energy mechanism of injury (e.g. motor vehicle accident, fall from height)
* Have an open fracture (i.e. the skin is broken at the fracture site), or
* Present with multiple injuries to the ipsilateral lower extremity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Grant, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baumgaertner MR, Curtin SL, Lindskog DM, Keggi JM. The value of the tip-apex distance in predicting failure of fixation of peritrochanteric fractures of the hip. J Bone Joint Surg Am. 1995 Jul;77(7):1058-64. doi: 10.2106/00004623-199507000-00012. PMID 7608228
- [Background] Lobo-Escolar A, Joven E, Iglesias D, Herrera A. Predictive factors for cutting-out in femoral intramedullary nailing. Injury. 2010 Dec;41(12):1312-6. doi: 10.1016/j.injury.2010.08.009. Epub 2010 Sep 15. PMID 20832795
- [Background] Geller JA, Saifi C, Morrison TA, Macaulay W. Tip-apex distance of intramedullary devices as a predictor of cut-out failure in the treatment of peritrochanteric elderly hip fractures. Int Orthop. 2010 Jun;34(5):719-22. doi: 10.1007/s00264-009-0837-7. Epub 2009 Jul 18. PMID 19618186
- [Background] De Bruijn K, den Hartog D, Tuinebreijer W, Roukema G. Reliability of predictors for screw cutout in intertrochanteric hip fractures. J Bone Joint Surg Am. 2012 Jul 18;94(14):1266-72. doi: 10.2106/JBJS.K.00357. PMID 22810396

RESULTS

PARTICIPANT FLOW:
Groups:
- ADAPT: Patients that receive intramedullary nail fixation with use of the ADAPT system
  Stryker ADAPT computer-assisted navigation: Adaptive Positioning Technology for Gamma 3
- Control: Patients that receive intramedullary nail fixation without use of the ADAPT system
Period: Overall Study
Arm/Group | ADAPT | Control
Started | 41 | 24
Completed | 26 | 24
Not Completed | 15 | 0
Not completed — First 12 patients were lead-ins | 12 | 0
Not completed — 3 consented screen fails | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ADAPT | Control | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 24 | 22 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 15 | 34
  Male | 7 | 9 | 16
Region of Enrollment [Number; unit: participants]
  United States | 26 | 24 | 50

OUTCOME MEASURES:

1. Primary Outcome: Tip-to-apex Distance
Description: Distance between lag screw tip and head surface as measured on the ADAPT system
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | ADAPT | Control
Number analyzed (Participants) | 26 | 24
mm | 14.1 (3.2) | 14.9 (3.0)

2. Secondary Outcome: Radiation Exposure
Description: Intraoperative fluoroscopy exposure time for lag screw placement (seconds)
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | ADAPT | Control
Number analyzed (Participants) | 26 | 24
seconds | 19.4 (8.8) | 18.8 (8.0)

ADVERSE EVENTS:
Time Frame: Start of surgery until end of surgery
Arm/Group | ADAPT | Control
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 0/26 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No